CLINICAL TRIAL: NCT02922751
Title: Childhood Liver Disease Research Network (ChiLDReN): FibroScan™ in Pediatric Cholestatic Liver Disease (FORCE) Study Protocol
Brief Title: FibroScan™ in Pediatric Cholestatic Liver Disease (FORCE)
Acronym: FORCE
Status: Completed | Type: Observational
Sponsor: Arbor Research Collaborative for Health (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: FORCE Study - ChiLDReN Network; U01DK103149 (NIH); U01DK103140 (NIH); U01DK103135 (NIH); U01DK084575 (NIH); U01DK084538 (NIH); U01DK084536 (NIH); U01DK062503 (NIH); U01DK062500 (NIH); U01DK062497 (NIH); U01DK062481 (NIH); U01DK062470 (NIH); U01DK062466 (NIH); U01DK062456 (NIH); U01DK062453 (NIH); U01DK062452 (NIH); U01DK062445 (NIH); U01DK062436 (NIH)
Record Dates: First submitted 2016-09-20; First posted 2016-10-04 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Biliary Atresia; Alagille Syndrome; Alpha1 Anti-Trypsin Deficiency; Portal Hypertension; Liver Fibrosis; Cholestasis
Keywords: transient elastography; pediatric liver disease; biliary atresia; Alagille Syndrome; Alpha1 Anti-Trypsin Deficiency; liver fibrosis; cholestasis
MeSH Terms: conditions — Biliary Atresia; Alagille Syndrome; alpha 1-Antitrypsin Deficiency; Hypertension, Portal; Liver Cirrhosis; Cholestasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- All Subjects: All subjects will be recruited from the Children parent studies: LOGIC (NCT00571272), BASIC (NCT00345553) and PROBE (NCT00061828) and will undergo Liver Stiffness Measurement (LSM). Subjects in these studies have one or more of the following conditions: biliary atresia (BA), Alpha1 Anti-trypsin Deficiency (A1AT) or Alagille Syndrome (ALGS).
  Interventions: Other: Liver Stiffness Measurement (LSM)

INTERVENTIONS:
Other: Liver Stiffness Measurement (LSM) — LSM will be measured via transient elastography utilizing the non-invasive FibroScan™ ultrasound device. LSM will be measured at Baseline, Year 1 and Year 2 visits.
  Other Names: FibroScan™

SUMMARY:
Noninvasive monitoring of liver fibrosis is an unmet need within the clinical management of pediatric chronic liver disease. While liver biopsy is often used in the initial diagnostic evaluation, subsequent biopsies are rarely performed because of inherent invasiveness and risks. This study will evaluate the role of non-invasive FibroScan™ technology to detect and quantify liver fibrosis.

DETAILED DESCRIPTION:
Noninvasive monitoring of liver fibrosis is an unmet and critical need within the clinical management of children with chronic liver disease. While liver biopsy is often used in the initial diagnostic evaluation of children with liver disease, subsequent surveillance liver biopsy is rarely performed in children because of its inherent invasiveness and risks. Therefore, our understanding of the natural history of fibrosis progression in children is limited. The patchy nature of fibrosis in many important pediatric liver diseases [e.g. biliary atresia (BA) and cystic fibrosis liver disease (CFLD)] limits the utility of sequential liver biopsy even if it were to be employed in clinical practice in pediatrics. Thus, non-invasive means of assessing liver fibrosis throughout the liver would be highly desirable and clinically useful in pediatric hepatology. ChiLDReN is poised and uniquely qualified to conduct a comprehensive longitudinal assessment of the utility of FibroScan™-specific elastography, liver stiffness measurement (LSM) as a measure of hepatic fibrosis in children with serious chronic cholestatic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 21 years at the time of enrollment
* Participants enrolled in a ChiLDReN based prospective observational cohort study (PROBE, BASIC, or LOGIC)
* Willingness and ability to participate in the study for up to 24 months
* One of the following three diagnoses

  * Biliary atresia per ChiLDReN criteria or,
  * Alpha-1 antitrypsin deficiency (PiZZ or SZ) or,
  * Alagille Syndrome per ChiLDReN criteria

Exclusion Criteria:

* BA with known situs inversus or polysplenia/asplenia
* Presence of clinically significant ascites detected on physical examination
* Open wound near expected FibroScan probe application site
* Use of implantable active medical device such as a pacemaker or defibrillator
* Known pregnancy
* Prior liver transplant
* Unable or unwilling to give informed consent or assent

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All children with an established diagnosis of BA (excluding those with known situs inversus or polysplenia/asplenia), who are actively followed at participating ChiLDReN sites and enrolled in PROBE or BASIC will be eligible for the trial. In addition, all children with A1AT or ALGS actively followed at one of these sites and enrolled in LOGIC will also be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Actual)
Dates: Start 2016-11-16 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Compare the distribution of LSM at enrollment between participants with and without portal hypertension | Enrollment
  A linear model will be fit to FibroScan™ values at enrollment to assess the impact of portal hypertension on LSM, controlling for important covariates such as age, gender, and race

SECONDARY OUTCOMES:
Change in Liver Stiffness Measurement (LSM) obtained via transient elastography from baseline to LSM at the Year 1 and Year 2 visits in participants with biliary atresia (BA). | Baseline, Year 1 Visit, Year 2 Visit
  The key secondary aim (Aim 2) compares the one- and two-year FibroScan™ values to those at enrollment in participants with BA.
Number of participants in whom a valid FibroScan™ LSM can be obtained | Baseline, Year 1 Visit, Year 2 Visit
  The investigators will define two measures of the feasibility of FibroScans™ in the participant populations with a "technically possible" FibroScan™, defined as the number of subjects with at least 10 FibroScan™ measurements obtained divided by the number assessed. The proportion of subjects with FibroScans™ of "acceptable quality" is defined as the number of subjects with FibroScan™ LSM with the ratio of the interquartile range and median of the 10 measurements <30%, of which at least 6 are completed, divided by the number assessed. The proportions and their 95% confidence intervals will be provided using the Wald method; however, the Wilson-Score methods will be used if the sample sizes are small or the proportion is small for a disease group. We will perform separate analyses for subjects <2 years of age and for those >2 years of age.
FibroScan™ LSM values at enrollment and conventional laboratory determinants of liver disease ((Pediatric End Stage Liver Disease (PELD) and APRI (Aspartate Aminotransferase (AST) to Platelet Ratio Index)). | Baseline
  The analysis will be limited to subjects for whom a PELD can be calculated (i.e., those for whom the individual components of the PELD score are available). Note that PELD will be calculated for all pediatric participants including those greater than 12 years of age. PELD is calculated as
  PELD = 4.80 x [ln serum bilirubin (mg/dL)] + 18.57 x [ln INR] - 6.87 x [ln albumin (g/dL)]
  + 4.36(<1 year old) + 6.67(growth failure) [www.unos.org]
  APRI is calculated as
  APRI = AST/upper limit of normal AST x 100 [U/L] Platelet Count (109/L) [U/L])

OTHER OUTCOMES:
Change from LSM Measurement obtained via transient elastography from baseline, to LSM at the Year 1 and Year 2 visits in participants with A1AT and ALGS | Baseline, Year 1, and Year 2 Visits in children with A2AT, ALGS, and BA.
  To prospectively explore changes in LSM over time by FibroScan™ in children with A1AT and ALGS.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Shneider, MD, Principal Investigator — Baylor College of Medicine; Ed Doo, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); Averell Sherker, MD, Study Director — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK); John Magee, MD, Principal Investigator — University of Michigan Medical Center, Ann Arbor; Lisa Henn, PhD, Principal Investigator — Arbor Research Collaborative of Health
Locations (13):
- United States (12):
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of California at San Francisco (UCSF), San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta (Emory University), Atlanta, Georgia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Cincinnati Children's Memorial Hospital, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Hospital (Baylor College of Medicine), Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared via the NIDDK's Data Repository.

REFERENCES:
- [Background] Pinzani M, Macias-Barragan J. Update on the pathophysiology of liver fibrosis. Expert Rev Gastroenterol Hepatol. 2010 Aug;4(4):459-72. doi: 10.1586/egh.10.47. PMID 20678019
- [Background] Trautwein C, Friedman SL, Schuppan D, Pinzani M. Hepatic fibrosis: Concept to treatment. J Hepatol. 2015 Apr;62(1 Suppl):S15-24. doi: 10.1016/j.jhep.2015.02.039. PMID 25920084
- [Background] Shneider BL, Abel B, Haber B, Karpen SJ, Magee JC, Romero R, Schwarz K, Bass LM, Kerkar N, Miethke AG, Rosenthal P, Turmelle Y, Robuck PR, Sokol RJ; Childhood Liver Disease Research and Education Network. Portal hypertension in children and young adults with biliary atresia. J Pediatr Gastroenterol Nutr. 2012 Nov;55(5):567-73. doi: 10.1097/MPG.0b013e31826eb0cf. PMID 22903006
- [Background] Teckman JH, Rosenthal P, Abel R, Bass LM, Michail S, Murray KF, Rudnick DA, Thomas DW, Spino C, Arnon R, Hertel PM, Heubi J, Kamath BM, Karnsakul W, Loomes KM, Magee JC, Molleston JP, Romero R, Shneider BL, Sherker AH, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Baseline Analysis of a Young alpha-1-Antitrypsin Deficiency Liver Disease Cohort Reveals Frequent Portal Hypertension. J Pediatr Gastroenterol Nutr. 2015 Jul;61(1):94-101. doi: 10.1097/MPG.0000000000000753. PMID 25651489
- [Background] Bonis PA, Friedman SL, Kaplan MM. Is liver fibrosis reversible? N Engl J Med. 2001 Feb 8;344(6):452-4. doi: 10.1056/NEJM200102083440610. No abstract available. PMID 11172184
- [Background] Ozaslan E. Drug-induced autoimmune hepatitis: an easily reversible type of liver fibrosis? Hepatology. 2011 Jan;53(1):370. doi: 10.1002/hep.23858. Epub 2010 Jul 29. No abstract available. PMID 20848612
- [Background] Saleh HA, Abu-Rashed AH. Liver biopsy remains the gold standard for evaluation of chronic hepatitis and fibrosis. J Gastrointestin Liver Dis. 2007 Dec;16(4):425-6. No abstract available. PMID 18193125
- [Background] Huang JF, Hsieh MY, Dai CY, Hou NJ, Lee LP, Lin ZY, Chen SC, Wang LY, Hsieh MY, Chang WY, Yu ML, Chuang WL. The incidence and risks of liver biopsy in non-cirrhotic patients: An evaluation of 3806 biopsies. Gut. 2007 May;56(5):736-7. doi: 10.1136/gut.2006.115410. No abstract available. PMID 17440193
- [Background] Falck-Ytter Y, McCullough AJ. The risks of percutaneous liver biopsy. Hepatology. 2001 Mar;33(3):764. doi: 10.1053/jhep.2001.0103303le01. No abstract available. PMID 11230761
- [Background] Westheim BH, Ostensen AB, Aagenaes I, Sanengen T, Almaas R. Evaluation of risk factors for bleeding after liver biopsy in children. J Pediatr Gastroenterol Nutr. 2012 Jul;55(1):82-7. doi: 10.1097/MPG.0b013e318249c12a. PMID 22249806
- [Background] El-Shabrawi MH, El-Karaksy HM, Okahsa SH, Kamal NM, El-Batran G, Badr KA. Outpatient blind percutaneous liver biopsy in infants and children: is it safe? Saudi J Gastroenterol. 2012 Jan-Feb;18(1):26-33. doi: 10.4103/1319-3767.91735. PMID 22249089
- [Background] Lachaux A, Le Gall C, Chambon M, Regnier F, Loras-Duclaux I, Bouvier R, Pinzaru M, Stamm D, Hermier M. Complications of percutaneous liver biopsy in infants and children. Eur J Pediatr. 1995 Aug;154(8):621-3. doi: 10.1007/BF02079063. PMID 7588960
- [Background] Castera L, Bernard PH, Le Bail B, Foucher J, Trimoulet P, Merrouche W, Couzigou P, de Ledinghen V. Transient elastography and biomarkers for liver fibrosis assessment and follow-up of inactive hepatitis B carriers. Aliment Pharmacol Ther. 2011 Feb;33(4):455-65. doi: 10.1111/j.1365-2036.2010.04547.x. PMID 21235598
- [Background] Kim S, Kang Y, Lee MJ, Kim MJ, Han SJ, Koh H. Points to be considered when applying FibroScan S probe in children with biliary atresia. J Pediatr Gastroenterol Nutr. 2014 Nov;59(5):624-8. doi: 10.1097/MPG.0000000000000489. PMID 25003372
- See also: Childhood Liver Disease Research Network (ChiLDReN) website — https://childrennetwork.org

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02922751/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/51/NCT02922751/ICF_000.pdf